CLINICAL TRIAL: NCT07280481
Title: Weekly Dynamics of Psychopathological and Symptom Networks During Mindfulness-Based Interventions for Emotional Distress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Associate Dean, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20251101
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Depression, Anxiety; Emotional Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIED group (Experimental): The experimental group will participate in a self-guided mindfulness-based intervention for emotional distress, delivered via a WeChat Mini Program platform. The intervention requires daily completion of learning modules and practice exercises. Psychological assessments utilizing self-report questionnaires will be conducted at: baseline (pre-intervention), weekly during the intervention phase (weeks 2 through 7), immediately post-intervention, and at the 1-month follow-up.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress (self-guided version)
- Waitlist control group (No Intervention): Participants in the waitlist control group will be offered access to the self-guided mindfulness-based intervention after completing all ten assessments (same as the experimental group).

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress (self-guided version) — The self-guided version of the Mindfulness Intervention for Emotional Distress (MIED) is a WeChat mini-program that lasts for 49 days. Each day, participants received different materials including (a) an audio recording of mindfulness meditation guidance; (b) learning materials in text or audio; and (c) assignments (for example, informal mindfulness practice, emotion journal, and challenging tasks). These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: MIED group

SUMMARY:
The goal of this clinical study is to learn how Mindfulness Intervention for Emotional Distress (MIED) helps people with emotional distress and how their symptoms and psychological patterns change over time.

The main questions it aims to answer are:

* How do the relationships between emotions, thoughts, and behaviors change week by week during mindfulness training?
* Which psychological skills, such as distress tolerance or cognitive flexibility, improve first and lead to later emotional relief? Two groups will be compared - one that takes part in an online mindfulness intervention and one that waits to join - to see how the intervention changes emotional and psychological networks over time.

Participants will:

* Complete a 7-week online self-guided Mindfulness Intervention for Emotional Distress（iMIED） designed for people experiencing high emotional distress.
* Fill out short weekly questionnaires about their emotions, thoughts, and behaviors before, during, and after the course (9 times in total).
* Receive access to the mindfulness program after the study if they are in the wait-list group.

This study includes about 500 adults aged 18 and older who feel anxious, depressed, or emotionally distressed but have no major psychiatric disorders. By tracking weekly changes, the research aims to identify how mindfulness intervention leads to emotional improvement and which skills play the most important roles in that process.

DETAILED DESCRIPTION:
Research Background Traditional psychotherapy research tends to emphasize description rather than explanation, relying excessively on data accumulation while neglecting theoretical construction and development (Gelo & Salvatore, 2016). Complex network theory and its related methods can overcome the limitations of traditional empiricism, providing a deeper theoretical framework and analytical tools for psychotherapy research. By applying complex network methods, it becomes possible to comprehensively analyze the multidimensional and multicausal dynamic relationships between symptoms or psychological variables during psychotherapy, thus gaining a clearer understanding of the processes underlying the development and recovery of mental health problems.

Network analysis can reveal the direct connections between different variables (Borsboom, 2017), rather than relying solely on changes in overall mean levels. Combined with multi-time-point measurement designs, researchers can track gradual changes in relationships between variables during the intervention, thereby identifying which associations change first in the therapeutic process and which variables may play key roles throughout the intervention (Blanken et al., 2019; Cervin et al., 2020). This contributes to an in-depth exploration of the mechanisms underlying psychological interventions and a more comprehensive understanding of change patterns in the therapeutic process.

Mindfulness-Based Interventions (MBIs) are a form of psychotherapy whose effectiveness has been widely validated (Wielgosz et al., 2019). Through regular mindfulness practice, individuals tend to develop healthier behavioral patterns, such as reduction of substance abuse, self-harm, suicidal behaviors, and eating disorder symptoms (Schuman-Olivier et al., 2020). Mindfulness-centered interventions are applicable to both clinical and non-clinical populations: not only to patients with physical or mental disorders (Carlson, 2012; Turgon et al., 2019), but also to individuals experiencing behavioral or emotional distress (Ju, 2022; Ma et al., 2018), all of whom can benefit from short-term or long-term mindfulness practice. Both traditional face-to-face formats and online mindfulness programs have been shown to improve emotional well-being and enhance quality of life (Li et al., 2025; Taylor et al., 2021). The convenience and accessibility of online interventions, in particular, enable more people experiencing emotional distress to receive continuous psychological support.

In addition to studying the efficacy of interventions, understanding the mechanisms of mindfulness interventions is equally important. Many researchers have begun to explore the mechanisms underlying Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy (MBCT) (Gu et al., 2015; Maloney et al., 2024). Traditional mechanism studies are mostly based on mediation models that conceptualize mechanisms as static variables linking interventions and outcomes (Kazdin, 2007), making it difficult to capture the dynamic interactions among multiple variables (such as distress tolerance, experiential avoidance, and cognitive flexibility) during the intervention process. The cross-diagnostic interactions and longitudinal predictive relationships between these transdiagnostic factors and anxiety or depressive symptoms during intervention remain unclear.

Therefore, to gain a deeper understanding of how mindfulness interventions "take effect" and the "change patterns" that occur during the process, this study is based on Liu's (2024) Rhombus Model of Psychopathology in Emotional Distress. Using a randomized controlled trial design, weekly measurements will be conducted on individuals participating in an online mindfulness intervention. By applying network analysis methods, this study will focus on the weekly dynamics of psychopathological and symptom networks formed by key mechanism variables-distress tolerance, experiential avoidance, life engagement, and cognitive flexibility-as well as anxiety and depression symptoms during the intervention. The aim is to systematically reveal the dynamic processes and core pathways through which mindfulness interventions drive psychological change.

Summary and Outlook

Summary of current research on mindfulness programs and main findings:

1. Existing studies have shown that online mindfulness programs help alleviate stress, anxiety, depression, and other forms of emotional distress.
2. The mechanisms underlying online mindfulness programs remain unclear. Traditional mechanism studies cannot capture the multidimensional and multicausal interactions between mechanism and outcome variables, nor their temporal dynamics.
3. Network analysis and dynamic systems analysis methods have shown promising potential in clinical science.

Based on the above summary, the following issues need to be further explored:

1. How do the psychopathological networks formed by transdiagnostic factors and anxiety/depression symptoms evolve week by week during mindfulness intervention?
2. During different stages of the intervention, which mechanism variables change first, and which changes may predict later treatment effects? Research Objectives

Based on the above summary, the overall objective of this study is to reveal the weekly dynamic characteristics and key pathways of psychological mechanisms and symptom networks among individuals with emotional distress during mindfulness intervention. The specific objectives are as follows:

1. To construct a weekly psychopathological network model of the mindfulness intervention process, systematically depicting the structural relationships among distress tolerance, experiential avoidance, cognitive flexibility, life engagement, and anxiety and depression symptoms;
2. To identify key mechanism variables and their temporal effects during intervention, revealing which psychological mechanisms change first and subsequently lead to improvements in other variables or symptoms;
3. To compare differences in network structures across different stages of intervention, clarifying the evolving patterns of network connection strength and node centrality indicators during the process.

Research Design The participants in this study will be adults. Participants will be recruited voluntarily and screened based on questionnaires included in the informed consent process. Inclusion criteria: 18 years or older, experiencing emotional distress such as depression or anxiety (Kessler-10 score > 21), no prior experience with mindfulness meditation, no current self-harm or suicidal risk, no bipolar disorder or schizophrenia, no history of substance abuse, and no severe personal trauma history.

After being randomly assigned to an intervention group or a waitlist control group, participants in the intervention group will take part in the self-guided mindfulness intervention for emotional distress, with a total of ten assessments: before the intervention, after each week during the intervention, after the intervention, and one week after one month post-intervention. The questionnaires will include, but are not limited to, measures of mindfulness, distress tolerance, experiential avoidance, cognitive flexibility, life engagement, and emotional distress. The waitlist control group will be allowed to participate in the self-guided mindfulness intervention for emotional distress after completing the ten assessments.

Withdrawal criteria: failure to complete questionnaires for two consecutive times; failure to check in via the mini-program for seven consecutive days.

Participants

Sample size:

The intervention group will include five classes conducted simultaneously, with a maximum capacity of 250 participants.

The control group will include an equivalent number of 250 participants.

Measures:

Demographics, K10, PHQ-9, GAD-7, OASIS, ODSIS, FFMQ-SF, TTT, CFI, BEAQ, DTS, ELS, RNT (Repetitive Negative Thinking), CPSS-SF.

ELIGIBILITY:
Inclusion Criteria:

* experiencing emotional distress such as depression or anxiety (Kessler-10 score > 21)

Exclusion Criteria:

* prior experience with mindfulness meditation
* current self-harm or suicidal risk
* bipolar disorder or schizophrenia
* history of substance abuse
* severe personal trauma history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-11-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Weekly changes of Overall Depression Severity and Impairment | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Overall Anxiety Severity and Impairment | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Weekly changes of treating thoughts as thoughts | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The questionnaire has 1 dimension and contains 5 items on a five-point Likert scale (1=completely compliant, 5=completely non-compliant), with higher scores indicating higher ability to treat ideas as ideas.
Weekly changes of Cognitive flexibility | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  Cognitive flexibility Inventory is a self-reported questionnaire measuring Cognitive flexibility level.Scores range from 20 to 100, with higher scores indicating higher levels of Cognitive flexibility.
Weekly changes of Brief Experiential Avoidance | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  Chinese version of the Brief Experiential Avoidance Questionnaire is used to measure Experiential Avoidance.Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of Distress Tolerance | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  Distress Tolerance Scale is used to measure Distress Tolerance. Scores range from 5 to 75, with higher scores indicating higher levels of Distress Tolerance.
Weekly changes of engaging in everyday life | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  Self-developed scale assessing the extent to which individuals' daily engagement in life domains (such as work, social interactions, and leisure activities) is affected by physical and psychological discomfort. , 16 items, scores range from 0 to 64, with higher scores indicating higher levels of engaging in everyday life.

SECONDARY OUTCOMES:
Weekly changes of Psychological Distress | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Weekly changes of depression | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The Patient Health Questionnaire-9 (PHQ-9) measures the severity of depressive symptoms over the past two weeks. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Weekly changes of anxiety | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The Generalized Anxiety Disorder-7 (GAD-7) measures the severity of generalized anxiety symptoms over the past two weeks. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 21, with higher scores indicating greater severity of anxiety symptoms.
Changes of trait mindfulness | before the intervention, during weeks 4 and 6 of the intervention, immediately after the intervention, 1 month after the intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Weekly changes of Perseverative Thinking | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  Perseverative Thinking Questionnaire,16 items, scores range from 0 to 60, with higher scores indicating greater severity of repetitive negative thinking (RNT).
Weekly changes in perceived stress | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The Chinese version of the Perceived Stress Scale - Short Form (CPSS-SF) is a 4-item self-report questionnaire assessing how unpredictable, uncontrollable, and overloaded individuals find their lives. Each item is rated on a 5-point scale from 0 (never) to 4 (very often). Total scores range from 0 to 16, with higher scores indicating greater perceived stress.
weekly changes of Self-Compassion | before the intervention, weekly during weeks 2-7 of the intervention, immediately after the intervention, 1 month after the intervention
  The Self-Compassion Scale-Short Form is a self-reported questionnaire measuring the level of self-compassion. Scores range from 12 to 60, with higher scores indicating higher levels of self-compassion.

OTHER OUTCOMES:
Sensory Processing Sensitivity | before the intervention
  The Chinese version of the Highly Sensitive Person Scale (HSPS) is a self-reported questionnaire designed to measure an individual's level of Sensory Processing Sensitivity (SPS). The scale consists of 27 items, with total scores ranging from 27 to 135. Higher scores indicate a higher level of sensory processing sensitivity, meaning the individual's traits are more inclined towards being a "highly sensitive person."

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (1):
- Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: No